CLINICAL TRIAL: NCT06692296
Title: Studio Pilota Sull'Efficacia Della Pedana Stabilometrica Nel Trattamento Del Paziente Con Atassia di Friedreich
Brief Title: Efficacy of Stabilometric Platform to Improve Standing Balance in Patients With Friedreich's Ataxia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Eugenio Medea (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1129; CET ANV 2024-97 (Other: Comitato Etico Territoriale Area Nord Veneto)
Record Dates: First submitted 2024-11-14; First posted 2024-11-18 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Friedreich Ataxia
Keywords: randomized controlled trial; Friedreich Ataxia; balance; rehabilitation; training; stabilometric platform; ataxia; therapeutic exercise; standing balance; Scale for the assessment and rating of ataxia; six minute walking test; functional reach test; timed up and go; Friedreich ataxia rating scale
MeSH Terms: conditions — Friedreich Ataxia; Ataxia

STUDY DESIGN:
Intervention Model Description: A monocentric, open-label randomized controlled trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Platform Group (Experimental): Balance training including both conventional rehabilitation (24 sessions) and training over a stabilometric platform (20 sessions).
  Interventions: Behavioral: Balance training over stabilometric platform; Behavioral: Balance training by means of conventional rehabilitation
- Conventional Group (Active Comparator): Balance training including only conventional rehabilitation (44 sessions).
  Interventions: Behavioral: Balance training by means of conventional rehabilitation

INTERVENTIONS:
Behavioral: Balance training over stabilometric platform — The treatment using the stabilometric platform (a total of 20 sessions) generally includes an initial phase (approximately 5 minutes) of training and warm-up in "monitor" mode, during which the patient becomes familiar with the equipment. The patient then moves on to "training library" mode, which includes the following subcategories: (1) Stabilometric tracings in both static and dynamic phases (10 minutes); (2) Dexterity exercises in both static and dynamic phases (10 minutes); (3) Imbalance exercises in both static and dynamic phases (10 minutes).
  The goal during this phase is to increase the patient's stability limits and provoke balance reactions through load shifts in all directions. The session concludes with 10 minutes of TecnoBody Exergames, which help to automate the functions learned within a more complex activity.
  Other Names: PROKIN - PK252
  Arms: Platform Group
Behavioral: Balance training by means of conventional rehabilitation — Conventional rehabilitation to improve balance includes an initial phase of tissue mobilization, particularly of the foot structures (approximately 5 minutes per foot), in order to prepare them for the subsequent activation phase. This is followed by a phase focused on activating the anti-gravity muscles and aligning the trunk within the chosen setting (10 minutes). The treatment continues with balance training, both static and dynamic, load transfers, and dual-task exercises using external references (15 minutes). The session concludes with functional exercises relevant to the patient's daily life context (10 minutes).
  Other Names: balance training

SUMMARY:
The primary objective is to evaluate the potential effectiveness of an individualized intensive rehabilitation intervention using the "Prokin 252" stabilometric platform in the treatment of adolescent and adult patients with Friedreich's Ataxia. The secondary objective is to assess the retention of the rehabilitation treatment effects over time.

Enrolled patients will be randomized and assigned to one of two treatment groups for four weeks. Three assessments will be conducted for each patient: one before treatment (T0), one at the end of treatment (T1), and a follow-up assessment 90 days after T1 via telemedicine (T2).

This study is:

* Exploratory: The study aims to explore the usefulness of the stabilometric platform in a rehabilitative setting in combination with conventional therapy;
* Not "first-in-human";
* Longitudinal: The study will investigate changes over time in motor and functional ability scales, as well as stabilometric platform parameters, within the same cohort;
* Randomized, controlled, open-label;
* Monocentric: The study will be conducted only at the "La Nostra Famiglia" Association in Conegliano and Pieve di Soligo - IRCCS Eugenio Medea in Conegliano - UOC Neuromotor Rehabilitation in Pieve di Soligo, Via Monte Grappa, 96, 31053 Pieve di Soligo TV;
* Prospective;
* Post-market.

DETAILED DESCRIPTION:
In recent years, there has been increasing interest in the scientific literature on degenerative diseases such as ataxic syndromes. Friedreich's Ataxia is one of the most common forms of hereditary ataxia. It is defined as a multisystemic neurodegenerative disorder with an autosomal recessive inheritance pattern, presenting both neurological and non-neurological clinical manifestations. The disease results from a mutation in the X25 gene on chromosome 9, characterized by an excessive repetition of the GAA trinucleotide, which leads to a reduction and malfunction of frataxin. Friedreich's Ataxia typically manifests in the first or second decade of life, with a significant functional impact and progressive disability. Often, initial symptoms are characterized by severe balance and coordination impairments, which not only affect functional independence but also patients' quality of life.

Currently, therapeutic options are very limited. Omaveloxolone is the first and only drug approved in 2023 by the Food and Drug Administration and The European Medicines Agency for adults and adolescents aged ≥16 with Friedreich's Ataxia. It has been shown to improve the score on the Modified Friedreich's Ataxia Rating Scale after chronic treatment. Rehabilitation is defined by the World Health Organization as a set of interventions designed to reduce disability and optimize functioning in individuals interacting with their environment. Current literature suggests that rehabilitation plays a central role in the treatment of Friedreich's Ataxia. Impairments and limitations associated with Friedreich's Ataxia can be addressed through rehabilitative procedures that, although they do not affect disease progression, may significantly improve the patient's functionality. Several studies indicated that the use of technological aids in neurorehabilitation leads to improvements in various conditions. Technological aids offer several advantages over traditional rehabilitation by significantly contributing to motor learning and brain plasticity, both of which are key to improving motor recovery. These aids can be easily tailored to the specific needs of each patient. Technology-based rehabilitation platforms can adjust the difficulty level and type of exercises according to the patient's progress, ensuring a personalized approach. The use of technologies such as virtual reality and interactive games makes rehabilitation more engaging and enjoyable. This increases patients' motivation to actively participate in rehabilitation sessions, improving adherence to treatment. Technologies can provide real-time feedback on patient performance, enabling immediate adjustments and enhancing motor learning. This type of feedback is crucial for improving body awareness and movement precision. Additionally, technologies can integrate visual, auditory, and tactile stimuli, which can enhance learning and brain plasticity.

One technological aid used in rehabilitation is the stabilometric platform. This consists of a platform equipped with sensors that record the oscillations of the body's center of gravity while the patient stands on it. These data can be used to analyze postural stability, detect balance problems, and monitor progress in rehabilitation programs. It is often used in fields such as physiotherapy, sports, and biomechanical research. In recent years, it has also been used as a rehabilitative tool to improve balance, coordination, and proprioception, including in the neurological field. Integrating the stabilometric platform into rehabilitation programs offers a more comprehensive and targeted approach to addressing balance and postural stability issues. Several studies have compared conventional rehabilitation with combined treatments involving the stabilometric platform. Results indicate that conventional balance training can improve balance function in patients, but when combined with visual feedback balance training, the improvements are more significant. In the literature, the use of the stabilometric platform combined with traditional physiotherapy has shown considerable effectiveness in resolving balance deficits in patients with various neurological conditions, though this has not been demonstrated in . In the literature on Friedreich's Ataxia, several studies have used this tool for assessment purposes. Balance parameters obtained using the stabilometric platform have shown a significant increase over time in patients with Friedreich's Ataxia, indicating impaired postural stability and balance while standing. These measures are significantly correlated with performance scores on the Friedreich's Ataxia Rating Scale, particularly with the Friedreich's Ataxia Rating Scale subscale on Upright Stability. However, there are no specific studies regarding the application of this device as a rehabilitative tool in Friedreich's Ataxia.

According to the existing literature, the investigators propose an open-label, monocentric, randomized pilot study to compare the effectiveness of a conventional rehabilitation program combined with training on the stabilometric platform (Group A) versus conventional rehabilitation alone (Group B) in improving balance reactions specifically in patients with mild to moderate Friedreich's Ataxia. The investigators will use the Prokin 252 system on the Tecnobody stabilometric platform. Enrolled patients will be randomly assigned to one of the two treatment groups for four weeks. Three assessments will be conducted for each patient: one before treatment (T0), one at the end of treatment (T1), and a follow-up assessment 90 days after T1 via telemedicine (T2). At T0 and T1, assessments will include tests and scales that measure the patient's overall functioning, commonly used in clinical practice, such as the Modified Friedreich's Ataxia Rating Scale, Scale for Assessment and Rating of Ataxia, 6-Minute Walk Test, Timed Up and Go, Berg Balance Scale, and Functional Reach Test. Additionally, using the stabilometric platform, patients will perform static stability and limits of stability tests while standing. At T2, patients will be reassessed via telemedicine with only the Modified Friedreich's Ataxia Rating Scale administered and Scale for Assessment and Rating of Ataxia. Changes in scores obtained on scales and on stabilometric platform parameters will serve as the evaluation criteria for the potential effectiveness of the treatment, also compared to the outcomes of standard physiotherapy treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 14 years;
* Weight < 150 kg;
* Genetic diagnosis of Friedreich's Ataxia;
* Subscores of SARA (Scale for the Assessment and Rating of Ataxia) as follows: (1) from 1 to 6 for the item 'Gait (walking ability)'; (2) from 1 to 3 for the item 'Stance (ability to maintain a stable posture)'; (3) ability to walk ≥10 metres with or without walking aids; (4) ability to stand unsupported; Stadiation of the Friedreich Ataxia Rating Scale between 2 and 4.

Exclusion Criteria:

* Age < 14 years;
* Diagnosis of acquired ataxia;
* Subscores for items on the SARA scale of: (1) 0 or 7 for gait; (2) 0 or 4-6 for stance;
* Inability to walk;
* Ability to walk < 10 meters;
* Standing position possible only with support;
* Other associated neurological conditions;
* Current major psychiatric disorder (psychosis and major depression).

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-02-03 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Score on the subscale 'Section E. Upright stability' of the modified Friedreich Ataxia Rating Scale. | Enrolment (T0), end of treatment at four weeks (T1), follow-up at 12 weeks after T1 (T2).
  The outcome evaluates balance performance while sitting, standing, and walking. Lower scores indicate better balance performance, higher scores indicate more severe balance impairment.

SECONDARY OUTCOMES:
Modified Friedreich's Ataxia Rating Scale (mFARS) | Enrolment (T0), end of treatment at four weeks (T1), follow-up at 12 weeks after T1 (T2).
  Clinical assessment of severity for neurological deficits, specifically designed for patients affected by Friedreich's Ataxia. The maximum score is 93, with higher scores indicating more severe neurological deficit. mFARS includes four subscales, evaluating 'bulbar' function (cough and speech), upper limb coordination, lower limb coordination, and upright stability (sitting, standing, walking).
Scale for Assessment and Rating for Ataxia (SARA). | Enrolment (T0), end of treatment at four weeks (T1), follow-up at 12 weeks after T1 (T2)..
  SARA is a semi-quantitative clinical assessment of cerebellar ataxia. It is composed by eight items: gait, stance, sitting, speech disturbance, finger chase, nose-finger test, fast alternating hand movements, heel shin slide. The final score ranges from zero (absence of ataxia) to 40 (severe ataxia).
Six minutes walking test (6MWT). | Enrolment (T0), end of treatment at four weeks (T1).
  6MWT is a clinical assessment of gait endurance, by measuring the distance covered (metres) while walking on a straight even path (30 meters) for six minutes. According to original instructions, the patient is asked to walk along the path as fast as possible, taking turns at the edges of the path. Patients are allowed to walk autonomously or with assistive devices and to rest by standing.
Timed Up and Go test (TUG). | Enrolment (T0), end of treatment at four weeks (T1).
  TUG evaluates mobility, balance, gait competence and fall risk. The test measures the time taken (seconds) to stand up from a standard armchair, walk three metres, turn and come back sitting. The patient cannot receive physical assistance during the test but is allowed to use assistive devices.
Berg balance scale (BBS). | Enrolment (T0), end of treatment at four weeks (T1).
  BBS is a clinical assessment of sitting balance, standing balance, and transfers. It's composed by 14 items, each item ranging from 0 (unable to complete the task) to 4 (able to complete the task according to time and instructions given). A higher score indicates better balance, with a score ≤43,5 predictive of fall risks.
Functional Reach Test (FRT). | Enrolment (T0), end of treatment at four weeks (T1).
  FRT evaluates dynamic balance while standing. Patient is asked to stand with one shoulder flexed at 90 degrees and the hand making a fist, and then to bend forward up to the limit of balance, right before taking a step to prevent falling. A horizontal ruler taped on the wall is used to measure the difference in position of the head of the third metacarpal bone from starting to end position. Patients are not allowed to touch the wall or rotate the trunk while bending forward.
Stabilometric platform. | Enrolment (T0), end of treatment at four weeks (T1).
  With the patient standing over a stabilometric platform, two kinematic assessments will be performed: (1) static stance, by standing for 30 seconds with eyes open and 30 seconds with eyes closed; (2) limits of stability, by bending with the body in different direction, displacing the centre of mass towards anterior, posterior, and lateral targets projected on a screen in front of the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriella Paparella, Medical Degree, Principal Investigator — Scientific Institute, IRCCS E. Medea, Department of Conegliano, Treviso, Italy.
Locations (1):
- Scientific Institute, IRCCS E. Medea, Department of Pieve di Soligo, Treviso, Italy, Pieve di Soligo, Veneto, Italy

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant data will be shared with other researchers upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Start date: January 2028; End date: January 2038.
Access Criteria: Any researcher accredited by non-profit clinical and research centre.

REFERENCES:
- [Background] Zesiewicz TA, Stephenson JB, Kim SH, Sullivan KL, Jahan I, Huang Y, Salemi JL, Wecker L, Shaw JD, Gooch CL. Longitudinal gait and balance decline in Friedreich's Ataxia: A pilot study. Gait Posture. 2017 Jun;55:25-30. doi: 10.1016/j.gaitpost.2017.03.019. Epub 2017 Mar 30. PMID 28411441
- [Background] Prosperini L, Pozzilli C. The clinical relevance of force platform measures in multiple sclerosis: a review. Mult Scler Int. 2013;2013:756564. doi: 10.1155/2013/756564. Epub 2013 May 19. PMID 23766910
- [Background] Podsiadlo D, Richardson S. The timed "Up & Go": a test of basic functional mobility for frail elderly persons. J Am Geriatr Soc. 1991 Feb;39(2):142-8. doi: 10.1111/j.1532-5415.1991.tb01616.x. PMID 1991946
- [Background] Milne SC, Kim SH, Murphy A, Larkindale J, Farmer J, Malapira R, Danoudis M, Shaw J, Ramakrishnan T, Rasouli F, Yiu EM, Georgiou-Karistianis N, Tai G, Zesiewicz T, Delatycki MB, Corben LA. The Responsiveness of Gait and Balance Outcomes to Disease Progression in Friedreich Ataxia. Cerebellum. 2022 Dec;21(6):963-975. doi: 10.1007/s12311-021-01348-2. Epub 2021 Dec 2. PMID 34855135
- [Background] Milne SC, Corben LA, Georgiou-Karistianis N, Delatycki MB, Yiu EM. Rehabilitation for Individuals With Genetic Degenerative Ataxia: A Systematic Review. Neurorehabil Neural Repair. 2017 Jul;31(7):609-622. doi: 10.1177/1545968317712469. Epub 2017 Jun 9. PMID 28595509
- [Background] Januario F, Campos I, Amaral C. Rehabilitation of postural stability in ataxic/hemiplegic patients after stroke. Disabil Rehabil. 2010;32(21):1775-9. doi: 10.3109/09638281003734433. PMID 20350209
- [Background] Ilg W, Milne S, Schmitz-Hubsch T, Alcock L, Beichert L, Bertini E, Mohamed Ibrahim N, Dawes H, Gomez CM, Hanagasi H, Kinnunen KM, Minnerop M, Nemeth AH, Newman J, Ng YS, Rentz C, Samanci B, Shah VV, Summa S, Vasco G, McNames J, Horak FB; Ataxia Global Initiative (AGI) working group Digital Motor Biomarkers. Quantitative Gait and Balance Outcomes for Ataxia Trials: Consensus Recommendations by the Ataxia Global Initiative Working Group on Digital-Motor Biomarkers. Cerebellum. 2024 Aug;23(4):1566-1592. doi: 10.1007/s12311-023-01625-2. Epub 2023 Nov 13. PMID 37955812
- [Background] Hartley H, Cassidy E, Bunn L, Kumar R, Pizer B, Lane S, Carter B. Exercise and Physical Therapy Interventions for Children with Ataxia: A Systematic Review. Cerebellum. 2019 Oct;18(5):951-968. doi: 10.1007/s12311-019-01063-z. PMID 31392562
- [Background] Cattaneo D, Jonsdottir J, Regola A, Carabalona R. Stabilometric assessment of context dependent balance recovery in persons with multiple sclerosis: a randomized controlled study. J Neuroeng Rehabil. 2014 Jun 10;11:100. doi: 10.1186/1743-0003-11-100. PMID 24912561
- [Background] Burciu RG, Fritsche N, Granert O, Schmitz L, Sponemann N, Konczak J, Theysohn N, Gerwig M, van Eimeren T, Timmann D. Brain changes associated with postural training in patients with cerebellar degeneration: a voxel-based morphometry study. J Neurosci. 2013 Mar 6;33(10):4594-604. doi: 10.1523/JNEUROSCI.3381-12.2013. PMID 23467375
- [Background] Bidichandani SI, Delatycki MB. Friedreich Ataxia. In: Adam MP, Pagon RA, Bird TD, Dolan CR, Stephens K, eds. GeneReviews™. Seattle: University of Washington; 2017.
- [Background] Berg K, Wood-Dauphinee S, Williams JI. The Balance Scale: reliability assessment with elderly residents and patients with an acute stroke. Scand J Rehabil Med. 1995 Mar;27(1):27-36. PMID 7792547